CLINICAL TRIAL: NCT02282384
Title: A Randomized Controlled Trial of Oseltamivir in Outpatients With Chronic Pulmonary Disease: a Pilot Study
Brief Title: An RCT of Oseltamivir in Outpatients With CPD: A Pilot Study.
Acronym: AVT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sites were unable to recruit participants
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AVT-2014
Record Dates: First submitted 2014-09-02; First posted 2014-11-04 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Disease; Influenza
MeSH Terms: conditions — Lung Diseases; Influenza, Human | interventions — Oseltamivir; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- oseltamivir (Experimental): 75 mg oseltamivir orally twice daily for 5 days within 72 hours of symptom onset
  Interventions: Drug: oseltamivir
- Placebo (Placebo Comparator): 75mg placebo calcium carbonate pills taken twice daily for five days within 72 hours of symptom onset and will be identical in appearance to oseltamivir
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: oseltamivir — They will be assessed for eligibility at the clinics and those randomized to the intervention will receive oseltamivir 75 mg orally twice daily for 5 days within 72 hours of symptom onset. Participants randomized to the control group will receive calcium carbonate placebo pills twice daily for five days within 72 hours of symptom onset. For patients with a known creatinine clearance < 10 ml/min, the recommended dose of 75mg orally daily for 5 days of either intervention or placebo will be administered.
  Other Names: Tamiflu
  Arms: oseltamivir
Other: Placebo
  Other Names: Calcium Carbonate
  Arms: Placebo

SUMMARY:
The proposed pilot study will provide needed data to establish the feasibility of a conducting a large randomized controlled trial as to the effectiveness of the use of oseltamivir early in the course of influenza in outpatients with chronic pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinic patients with physician diagnosed chronic obstructive pulmonary disease
* respirologist-diagnosed non-cystic fibrosis bronchiectasis and pulmonary fibrosis (based on appropriate clinical, exposure, and radiological criteria as per American Thoracic Society guidelines)
* Participants will be drawn from the respirology clinics and will be randomized if within 72 hours of meeting criteria for influenza-like illness

Exclusion Criteria:

* residents of nursing homes
* patients who are immunosuppressed
* patients on immunosuppressive does (15 mg or more) of prednisone for three weeks or longer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
non-elective admission to hospital | up to 28 days following randomization
  A non-elective admission to hospital, in contrast to visits to the emergency department where admission does not take place. However, a prolonged stay in the emergency department (> 24 hours) will also be considered to be hospitalization. Events that occur beyond this time period are deemed unlikely to be directly related to influenza,except functional status which will be assessed up to three months following acute respiratory infection. Secondly, the hospitalization must also be considered to be due to acute respiratory illness. An adjudication committee (comprised of two infectious diseases physicians who also practice general internal medicine) blinded to study group allocation will review data for hospitalization. They will be asked to judge whether the hospitalization was definitely or probably related to the acute respiratory illness. Those judged to be definitely or probably related will be considered as our primary outcome.

SECONDARY OUTCOMES:
lower respiratory tract infection | up to 28 days following randomization
  lower respiratory tract infection including exacerbation of chronic pulmonary disease

OTHER OUTCOMES:
pneumonia | up to 28 days following randomization
neutrophilic bronchitis | up to 28 days following randomization
acute sinusitis | up to 28 days following randomization
antimicrobial prescriptions | up to 28 days following randomization
visits to medical providers | up to 28 days following randomization
  visits to emergency department without admission and non-routine visits to other physician clinics will be assessed separately
changes in functional status | up to 3 months from randomization
  This outcome will be measured using Activities of Daily Living (ADL) score, an index of independence of activities of daily living. Will be assessed at baseline, 2 weeks, 1 month, 3 months after acute respiratory infection onset
absenteeism from work | up to 28 days from randomization
additional care or support needed in the home | up to 3 months following randomization
  Need for new or additional informal caregiver support in the home, need for professional help in the home, transfer to a residential facility, need for rehabilitation for up to 3 months.
laboratory testing using RT-PCR for influenza | up to 28 days following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD, Principal Investigator — McMaster University